CLINICAL TRIAL: NCT01104207
Title: Clinical Trial of Transcranial Magnetic Stimulation for Relief of Tinnitus
Brief Title: Transcranial Magnetic Stimulation for Tinnitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: C7448-I
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Tinnitus
Keywords: tinnitus; TMS; transcranial magnetic stimulation
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Half of the study participants will receive 2000 pulses of 1 Hz active rTMS daily on 10 consecutive work days.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Arm 2 (Sham Comparator): Half of the study participants will receive 2000 pulses of 1 Hz placebo rTMS daily on 10 consecutive work days.
  Interventions: Device: placebo rTMS

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — rTMS involves application of electromagnetic pulses through a coil to the subject's scalp. Some of the electromagnetic energy is transmitted to underlying neural tissue. The goal for this study: 1 Hz rTMS will suppress neural activity responsible for tinnitus perception.
  Arms: Arm 1
Device: placebo rTMS — placebo rTMS
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess the effectiveness of repetitive transcranial magnetic stimulation (rTMS) for reducing the loudness or severity of chronic tinnitus.

DETAILED DESCRIPTION:
This is a prospective, randomized, subject and clinician/observer blind, placebo-controlled parallel-group clinical trial of rTMS involving people who experience chronic tinnitus. Eligible subjects are randomly assigned to receive either active rTMS treatment or placebo treatment to either the left or right side of the head. Subjects receive 2000 pulses of 1 Hz rTMS therapy daily on 10 consecutive work days. Outcomes are measured prior to the start of treatment and after the last therapeutic session. Follow-up evaluations are conducted 1, 2, 4, 13 and 26 weeks after the last treatment session. This design allows us to determine if rTMS reduces the severity and loudness of tinnitus, the long-term duration of relief, and whether the target for coil placement (left/right side of head) affects active rTMS efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic tinnitus.
* Able to provide written informed consent.
* Subject is naive regarding rTMS.
* Age/Gender: minimum 18 years old, with an attempt to sample equal numbers of male and female subjects.
* Other concurrent treatments: A four-week washout from any other tinnitus treatment or management program is required prior to entering this study.
* Other medications: No restrictions, provided the dosages have been in place for at least 6 months.
* Psychological status: Stable enough to complete this study per the opinion of the Study Physician.
* Hearing function: All degrees of hearing function can be included recognizing that profound, bilateral losses will not be able to perform tinnitus evaluations and hearing tests, but will be able to rate subjective tinnitus loudness, annoyance and impact on life. This is an important subpopulation because of the challenges in treating them with acoustic therapy and the need for a medical intervention.
* Tinnitus characteristics: All forms of tinnitus etiology will be accepted, providing the following criteria are met:

  * Tinnitus duration: Not less than 1 year. Cases of less than 1 year duration have increased likelihood of resolving spontaneously.
  * Stability: Constant (not pulsatile, intermittent, varying to a high degree in loudness or changing in location of perception). Fluctuating tinnitus reduces the reliability of test-retest measures for loudness.
  * Self-rated tinnitus loudness: >= 6 on a visual numerical scale (VNS: 0 labeled "No Tinnitus", 10 labeled "Very Loud"). This outcome measure will provide a subjective indication of immediate changes in perceived loudness.
  * Location of tinnitus perception: Unrestricted. Tinnitus may be unilateral, bilateral, or perceived in the head.

Exclusion Criteria:

* Medical conditions: No active neurologic or otologic disease processes that may impact tinnitus perception. No auto-immune diseases. No pregnancy or planned pregnancy during the study. No women who are lactating or are of child-bearing-age without using contraception.
* Objective Tinnitus - tinnitus that is audible to other people in addition to the patient. This type of tinnitus is rare and is unlikely to respond to rTMS because it is not associated with abnormal neural activity in the central auditory system.
* History or evidence of significant brain malformation or neoplasm, head injury, cerebral vascular events (such as strokes), neurodegenerative disorders affecting the brain (such as Parkinson's Disease, ALS, Huntington's Disease or Multiple Sclerosis) or prior brain surgery.
* Cardiac pace makers, other electronic implants (including cochlear implants), intracranial or intraocular metallic particles.
* History of seizures or epileptic activity.
* Patients who cannot communicate reliably with the investigator or who are not likely to cope with the requirements of the trial.
* Participation in a clinical trial within the last 30 days before the start of this one.
* Maximum number of previous clinical trials for tinnitus in which subjects may have participated: two.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Folmer, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Theodoroff SM, Griest SE, Folmer RL. Transcranial magnetic stimulation for tinnitus: using the Tinnitus Functional Index to predict benefit in a randomized controlled trial. Trials. 2017 Feb 9;18(1):64. doi: 10.1186/s13063-017-1807-9. PMID 28183355
- [Derived] Folmer RL, Theodoroff SM, Casiana L, Shi Y, Griest S, Vachhani J. Repetitive Transcranial Magnetic Stimulation Treatment for Chronic Tinnitus: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2015 Aug;141(8):716-22. doi: 10.1001/jamaoto.2015.1219. PMID 26181507

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: For half of the subjects, rTMS will be delivered to one side of the head.
  repetitive transcranial magnetic stimulation (rTMS): rTMS involves application of electromagnetic pulses through a coil to the subject's scalp. Some of the electromagnetic energy is transmitted to underlying neural tissue. The goal for this study: 1 Hz rTMS will suppress neural activity responsible for tinnitus perception.
- Arm 2: For half of the subjects, placebo rTMS will be delivered to one side of the head.
  placebo rTMS: placebo rTMS
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 35 | 35
Completed | 32 | 32
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 19 | 44
  >=65 years | 10 | 16 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.5) | 62.8 (8.3) | 60.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 28 | 28 | 56
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
Tinnitus Functional Index [Mean (Standard Deviation); unit: units on a scale] — The TFI is a 25-item questionnaire that assesses tinnitus severity. The possible range of scores for the TFI is 0 to 100, with higher scores indicating more severe tinnitus.
  units on a scale | 44.8 (19.4) | 40.6 (22.2) | 42.7 (20.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Tinnitus Functional Index (TFI) Score
Description: The TFI is a 25-item questionnaire that assesses tinnitus severity. The possible range of scores for the TFI is 0 to 100, with higher scores indicating more severe tinnitus.
Time Frame: 26 weeks post-treatment
Measure: Mean (Standard Deviation); unit: units on TFI scale; change from baseline
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 32 | 32
units on TFI scale; change from baseline | -13.8 (15.2) | -2.9 (15.8)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes